CLINICAL TRIAL: NCT02153697
Title: Comparative Study Investigating the Therapy of of Solar Lentigines With the Q-switched SINON Rubin 694nm Laser Versus Pigmanorm® Cream
Brief Title: Comparative Study of the Therapy of Solar Lentigines With a Q-switched Rubin Laser Versus a Bleaching Cream
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEK-ZH-Nr. 2013-0435
Record Dates: First submitted 2014-05-20; First posted 2014-06-03 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Solar Lentigines
Keywords: solar lentigines; Q-switches Laser; bleaching cream

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pigmanorm Cream, Q-switched Ruby laser,solar lentigines (Experimental): Solar lentigines on the left back of the hand side are treated with Pigmanorm Cream once a day for 7 weeks. Solar lentigines on the right back of the hand side are treated with a Q-switched Ruby laser at Baseline and if required at day 28.
  Interventions: Device: Q-switched SINON Ruby Laser; Drug: Pigmanorm Cream

INTERVENTIONS:
Device: Q-switched SINON Ruby Laser — Solar lentigines on the right back of the hand side are treated with the Q-switched SINON Ruby Laser at Baseline and if required at day 28.
Drug: Pigmanorm Cream — Solar lentigines on the left back of the hand side are treated once a day during 7 weeks with Pigmanorm cream, a bleaching cream containing hydrochinon.

SUMMARY:
Benign pigmented lesions as solar lentigines are a common finding in Caucasian individuals. Their removal may be requested for aesthetic reasons.

The goal of the study is comparing the efficacy and tolerance of two different therapy modalities established for treating solar lentigines.

The right back of the hand side will be treated with the Q-switched SINON Rubin 694nm Laser, the left back of the hand side with a hydrochinon containing bleaching cream (Pigmanorm® cream).

The investigators estimate that a physical therapy with a Q-switched Rubin laser system is more effective in the removal of solar lentigines than a topical chemical therapy with a hydrochinon containing bleaching cream.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50
* female patient must be in post-menopause (> 2 years)
* Clinically and dermoscopic confirmed solar lentigines on both sides back of the hands

Exclusion Criteria:

* non melanocytic pigmentation, vitiligo, melanoma and suspicion of melanoma
* intolerance against an ingredience of pigmanorm® cream
* acute inflammation or eczema on back of the hands
* patients with renal disease
* intake of photosensibilisating medication in the past 3 months
* treatment of solar lentigines on back of the hands in the past 6 months
* solarium or sun exposure about 6 weeks before and after treatment
* immunsuppressed patients

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of clearing of pigmentation | 140 days (Baseline, Day 28, Day 56, Day 140)
  The primary efficacy objective is to evaluate the clearing of pigmentation(percentage of clearing) following a quartile scale of poor (25% clearance), fair (26-50% clearance), good (51-75% clearance), and excellent (76-100% clearance).

SECONDARY OUTCOMES:
Evaluation of safety profile | 140 days (Baseline, Day 28, Day 56, Day 140)
  Adverse effects are noted at each visit.
Change from Baseline in Pigmentation at day 140 | Long term outcome is assessed 3 months after finishing treatment.
  The clearing of pigmentation (percentage of clearing) following a quartile scale of poor (25% clearance), fair (26-50% clearance), good (51-75% clearance), and excellent (76-100% clearance) is assessed at day 140 from Baseline ( = 3 months after finishing treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Division of Dermatology, Zurich, Switzerland